CLINICAL TRIAL: NCT06887660
Title: Speech-language Skills of Orthodontic Residents Through the Use of the "Interdisciplinary Orofacial Examination Protocol for Children and Adolescents": Single-group Pre-post Study With External Validation
Brief Title: Speech-language Skills of Orthodontic Residents Through the Use of the "Interdisciplinary Orofacial Examination Protocol for Children and Adolescents"
Status: Completed | Type: Observational
Sponsor: University of Pavia (Other)
Responsible Party: Principal Investigator, Andrea Scribante, Associate Professor, Principal Investigator, University of Pavia
Other Study IDs: 2025-SPEECHTHERAPY
Record Dates: First submitted 2025-03-09; First posted 2025-03-20 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Mouth Breathing
Keywords: Orthodontic diagnosis
MeSH Terms: conditions — Mouth Breathing

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Orthodontic patients: Orthodontic patients at their first dental visit
  Interventions: Other: Orthodontic diagnosis

INTERVENTIONS:
Other: Orthodontic diagnosis — Initial Assessment Orthodontic residents assessed each patient based on their existing knowledge of speech therapy. They rated the necessity for a speech therapy consultation on a scale from 1 to 10, with 1 indicating "not necessary" and 10 indicating "absolutely necessary."
  Protocol-Guided Assessment The same residents then reassessed the same patients using the Interdisciplinary Orofacial Evaluation Protocol. After this evaluation, they again rated the necessity for a speech therapy consultation using the same 1 to 10 scale.
  Speech-therapist Evaluation Subsequently, a speech therapy specialist independently evaluated each patient using the same protocol and provided their rating for the necessity of a speech therapy consultation on the same scale.

SUMMARY:
This single-group pre-post study with external validation will be conducted on 29 orthodontic residents at the University of Pavia to assess their ability to recognize orofacial myofunctional disorders (OMD) before and after using an Interdisciplinary Orofacial Examination Protocol for Children and Adolescents. Even though this was the main purpose, the study investigated also the effectiveness of the Protocol in guiding the diagnosis of OMD.

DETAILED DESCRIPTION:
This single-group pre-post study with external validation aims to investigate the knowledge of orthodontic residents in the diagnosis of OMD. The study will be conducted on a sample of 29 residents enrolled at the Postgraduate Program of Orthodontics of the University of Pavia. Parents/legal guardians will be asked to sign the informed consent for the participations of patients in the study. The study cohort will be constituted of orthodontic patients aged 6-18 that will be visited for their first time at the Unit of Orthodontics and Pediatric Dentistry, Section of Dentistry, Department of Clinical, Surgical, Diagnostic, and Pediatric Sciences of the University of Pavia.

The first part of the study will involve the administration to the parents of the patients an anamnestic form aimed to investigate the patient's general health status, potential oral habits, respiratory condition, and any speech disorders. The responses to the questionnaire will be categorized as "Yes," "No," or "Sometimes.". Following the completion of the questionnaire, orthodontic residents will be asked to evaluate the patients based on their current knowledge of speech therapy and to determine the necessity of a trained speech therapy consultation. They will record their assessments on a dedicated form, rating the necessity on a scale from 1 to 10, where 1 indicates no necessity and 10 indicates absolute necessity (T0). After this initial assessment, the same residents will reassess each patient using the Interdisciplinary Orofacial Examination Protocol as a guideline (T1). Once they will complete this second evaluation, they will be required to rate the necessity for speech therapy consultation on the same 1 to 10 scale. In the final step (T2), each patient will be evaluated after 2 weeks by a specialist speech therapist using the same protocol. The speech therapist will independently assign a final score from 1 to 10, indicating the necessity for further speech therapy evaluation. After all evaluations will be completed, the responses will be codified into a scoring system, allowing to quantify the severity of each dysfunction. The Interdisciplinary Protocol used in this study comprises 15 items designed to assess patients from orthodontic, myofunctional, and phonatory perspectives.

These includes the evaluation of facial profile, breathing pattern, nasal airway function, lip seal at rest, and different types of malocclusions, such as vertical, sagittal, and transverse.

The protocol also measures overbite, overjet, and dental alignment, along with tonsil hypertrophy, tongue mobility, swallowing function, and articulation of speech sounds.

Data will be statistically analysed with data normality assessment and appropriate parametric or non-parametric test (significance threshold: p<0.05).

ELIGIBILITY:
Inclusion Criteria:

* Patients at their first dental visit
* No previous orthodontic treatment.

Exclusion Criteria:

* Patients with history of orthodontic therapy
* Patients with history of speech therapy
* Patients presenting cranio-facial syndroms and malformations

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients scheduled for orthodontic evaluation will be visited for the first time at the Unit.
Sampling Method: Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2025-03-30 (Actual); Primary Completion 2025-06-04 (Actual); Study Completion 2025-06-10 (Actual)

PRIMARY OUTCOMES:
Change in Diagnostic score | Baseline and after 2 weeks
  Score from 0 to 10 of the speech-language treatment need indicated by the Orthodontic Resident and confirmed by the diagnosis of a calibrated speech-language therapist.

SECONDARY OUTCOMES:
Profile | Baseline and after 2 weeks
  It evaluates the patient's facial profile to identify any deviations from normal alignment. Classifications include normal, slightly concave/convex, or severely concave/convex profiles.
Respiration pattern | Baseline and after 2 weeks
  It assesses the patient's habitual breathing method, determining if it is nasal, mixed, or oral. This evaluation helps identify potential respiratory issues that may affect orofacial development.
Nostril Patency During Forced Breathing | Baseline and after 2 weeks
  It examines the degree of nasal airway obstruction during forced inhalation. Grades range from 0 (both nostrils dilate) to 5 (bilateral total collapse), providing insight into nasal airflow efficiency.
Lips at Rest | Baseline and after 2 weeks
  It observes the patient's lip posture to determine if a natural lip seal is present without effort, achieved with effort, or absent. This assessment is crucial for understanding lip function and potential impacts on oral health.
Vertical Malocclusion | Baseline and after 2 weeks
  It evaluates the vertical relationship between the upper and lower dental arches in maximum intercuspation. Classifications include normal occlusion, mild deep/open bite, or severe deep/open bite, indicating vertical alignment issues.
Sagittal Malocclusion | Baseline and after 2 weeks
  It assesses the anteroposterior relationship of the molars to classify occlusion as Class I (normal), moderate Class II/III, or complete Class II/III, identifying discrepancies in jaw alignment.
Transverse Malocclusion | Baseline and after 2 weeks
  It evaluates the transverse relationship between the dental arches, identifying normal alignment, edge-to-edge bite, or complete crossbite, which can affect chewing efficiency and facial symmetry.
Overbite | Baseline and after 2 weeks
  It measures the vertical overlap between the upper and lower incisors. A normal overbite ranges between 2 to 3 millimeters; deviations may be classified as slightly or severely increased/reduced, impacting esthetics and function.
Overjet | Baseline and after 2 weeks
  It assesses the horizontal distance between the upper and lower incisors. A normal overjet is 2 to 3 millimeters; variations can be slightly or severely increased/reduced, influencing speech and biting.
Dental Alignment | Baseline and after 2 weeks
  It observes for crowding or spacing (diastemas) in the dental arches. Classifications include normal alignment, mild crowding/spacing, or severe crowding/spacing, which can affect oral hygiene and occlusion.
Tonsil Size | Baseline and after 2 weeks
  It assesses the degree of tonsillar hypertrophy, ranging from Grade 0 (tonsillectomy) to Grade 5 (tonsils occupying more than 75% of the oropharynx), which can influence breathing and swallowing functions.
Lingual Mobility | Baseline and after 2 weeks
  It evaluates tongue mobility by asking the patient to touch the palate with the tongue tip. Grades range from 0 (post-frenulectomy) to 5 (tongue tip does not reach the lower incisor edge), identifying potential restrictions like tongue-tie.
Muscle effort during swallowing | Baseline and after 2 weeks
  It observes the perioral muscle activity during swallowing, noting absence of effort, slight effort, or excessive effort, which can indicate dysfunctional swallowing patterns.
Tongue movement during swallowing | Baseline and after 2 weeks
  It assesses tongue positioning during swallowing by having the patient hold and swallow a sip of water while the examiner observes for normal movement, anterior tongue thrust, or tongue interposition, which can affect dental alignment.
Speech articulation | Baseline and after 2 weeks
  It evaluates phoneme production by having the patient repeat specific Italian words (e.g., "tetto," "lalla," "ciuccio," "sasso," "stella," "ramarro," "zanzara"). Observations include adequate articulation, sound distortions, or omission of sounds, aiding in the identification of speech disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Scribante, DDS, PhD, Principal Investigator — University of Pavia
Locations (1):
- Unit of Orthodontics and Pediatric Dentistry - Section of Dentistry - Department of Clinical, Surgical, Diagnostic and Pediatrics - University of Pavia, Pavia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No
Data will be available upon motivated request to the Principal Investigator.